CLINICAL TRIAL: NCT03224637
Title: Fluoroscopic Guided Radiofrequency of Genicular Nerves for Pain Alleviation in Chronic Knee Osteoarthritis : A Single-blind Randomized Controlled Trial.
Brief Title: Radiofrequency Neurotomy In Relieving Chronic Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Lecturer of Anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00009913
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Osteo Arthritis Knee; Pain, Chronic
MeSH Terms: conditions — Chronic Pain | interventions — Acetaminophen; Congresses as Topic; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiofrequency group (Active Comparator): radiofrequency was done in the three genicular nerves upper medial and upper lateral and lower medial
  Interventions: Procedure: radiofrequency
- conventional group (Active Comparator): the patients received conventional paracetamol and non steroidal antiinflammatory
  Interventions: Drug: Paracetamol (conventional); Drug: Ketorolac Tromethamine (conventional)

INTERVENTIONS:
Procedure: radiofrequency — radiofrequency done in the three genicular nerves upper medial and upper lateral and lower medial
  Arms: radiofrequency group
Drug: Paracetamol (conventional)
  Arms: conventional group
Drug: Ketorolac Tromethamine (conventional)
  Arms: conventional group

SUMMARY:
Osteoarthritis (OA) affects aged above 45 years. RF has been used for several painful conditions. There have been a few attempts to use RF current for the treatment of painful conditions of joints of the extremities. It was also used for the treatment of painful conditions of the hip joint.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is commonest chronic arthritis affecting patients usually aged above 45 years. OA decreased health-related quality of life and increased economic costs. Radiofrequency (RF), was used for the treatment of chronic pain unresponsive to conservative therapies. RF has been used for several painful conditions. There have been a few attempts to use RF current for the treatment of painful conditions of joints of the extremities. It was also used for the treatment of painful conditions of the hip joint.

ELIGIBILITY:
Inclusion Criteria:

* chronic arthritis according to the American College of Rheumatology criteria
* diagnosed radiologically patients in stage 3 and 4, according to the Kellgren-Lawrence classification

Exclusion Criteria:

* other causes of pain such as radiculopathy, neurological disorders, or intermittent claudication.
* patients receive intraarticular steroid or hyaluronic acids during previous three months.
* patients did previous knee surgery.
* Patients with general contraindication to the application of invasive intervention such as hemorrhage, coagulation disorder, systemic infection or local infection.
* patients with other connective tissue disease affecting the knee. And 6-psychiatric disorders.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
pain assessment by VAS scale | 6 months
  assessing pain by VAS scale

SECONDARY OUTCOMES:
patient satisfaction by Likert scale | 6 months
  Likert scale to assess patients satisfaction
patient disability by Western Ontario McMaster Universities OA index | 6 months
  Western Ontario McMaster Universities OA index to assess disability

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] El-Hakeim EH, Elawamy A, Kamel EZ, Goma SH, Gamal RM, Ghandour AM, Osman AM, Morsy KM. Fluoroscopic Guided Radiofrequency of Genicular Nerves for Pain Alleviation in Chronic Knee Osteoarthritis: A Single-Blind Randomized Controlled Trial. Pain Physician. 2018 Mar;21(2):169-177. PMID 29565947